CLINICAL TRIAL: NCT00329576
Title: Evaluate the Anti-HBs Antibody Persistence, in Subjects Who Received GSK Biologicals' Preservative-free or Thiomersal-free Engerix™-B or Engerix™-B Containing Thiomersal, Approximately 5 to 6 Yrs Earlier
Brief Title: Evaluate Immune Response Approximately 5 to 6 Years After Receiving Different Formulations of GSK Bio Hep B Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 106640
Record Dates: First submitted 2006-05-23; First posted 2006-05-24 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

INTERVENTIONS:
Biological: Hepatitis B vaccine

SUMMARY:
To evaluate the persistence of antibodies against hepatitis B, approximately 5 to 6 years after the first dose of the hepatitis B in the primary vaccination study.

DETAILED DESCRIPTION:
All subjects who participated in the primary vaccination study, where subjects who received GSK Biologicals' hepatitis B vaccine and who will consent to participate in this long-term follow-up study, approximately 5 to 6 years after the primary vaccination study. The study will be conducted in only 3 centres out of the 4 centres in the primary vaccination study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have participated in the primary study and should have received the first primary dose of vaccination more than five years ago and less than six years ago before blood sampling in this long-term follow-up study.
* Written informed consent obtained from the subject for the long-term follow-up.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 632
Dates: Start 2006-05; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Wilrijk, Belgium
- GSK Investigational Site, Munich, Bavaria, Germany
- GSK Investigational Site, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Van Damme P, von Sonnenburg F, Hatz C, Hoet B, Lefevre I, Leyssen M. Long-term immunogenicity of preservative-free hepatitis B vaccine formulations in adults. J Med Virol. 2009 Oct;81(10):1710-5. doi: 10.1002/jmv.21568. PMID 19697416
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 106640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register